CLINICAL TRIAL: NCT02218398
Title: Bronchodilator Test in Mechanical Ventilated Chronic Obstructive Pulmonary Disease Patients, a Randomized Controlled Trial
Brief Title: Bronchodilator Test in Mechanical Ventilated Chronic Obstructive Pulmonary Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Jie Li, RRT-NPS, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BJCYRT-002
Record Dates: First submitted 2014-02-06; First posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: airway resistance; lung compliance; Duration of mechanical ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bronchodilator (Experimental): Albuterol 3-4 times per day, steroids when necessary.
  Interventions: Drug: Albuterol
- No drug (No Intervention): No drug

INTERVENTIONS:
Drug: Albuterol
  Arms: Bronchodilator

SUMMARY:
Investigators developed a test to assess the bronchodilator effects in mechanically ventilated chronic obstructive pulmonary disease patients by comparing the change of airway resistance. No matter whether patients respond to bronchodilator or not, they are randomized assigned to bronchodilator 3-4 times per day group and no bronchodilator group. Then investigators could objectively decide whether individual patients need or benefit from bronchodilator administration.

DETAILED DESCRIPTION:
Bronchodilator is commonly used in mechanical ventilated chronic obstructive pulmonary disease patients. It is assumed that patient's response to bronchodilator is the same during acute exacerbation or when stable whether on mechanical ventilation or not. Decision to treat is often independent of response and the patient's response to the medicine is not precisely evaluated. Investigators developed a test to assess the bronchodilator effects in mechanically ventilated chronic obstructive pulmonary disease patients by comparing the change of airway resistance. No matter whether patients respond to bronchodilator or not, they are randomized assigned to bronchodilator 3-4 times per day group and no bronchodilator group. Then investigators could objectively decide whether individual patients need or benefit from bronchodilator administration.

ELIGIBILITY:
Inclusion Criteria:

should meet all the criteria:

1. Acute exacerbated chronic obstructive pulmonary disease
2. Invasive mechanical ventilation with intubation outside ICU no more than 48 hours

Exclusion Criteria:

Meet any of the criteria:

1. Asthma
2. Tracheotomy
3. Prolonged Mechanical Ventilation (Have been mechanical ventilated for more than 21 days)
4. Unstable hemodynamic status
5. Severe pneumonia
6. Contraindication for bronchodilator
7. Contraindication for sedation
8. Refusal to participate in study
9. Re-intubation in 48 hours
10. Mental disorder, could not understand and accomplish pulmonary function test

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of 12% Decrease in airway resistance | 30 minutes

SECONDARY OUTCOMES:
Duration of mechanical ventilation | participants will be followed for the duration of ICU stay, an expected average of 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory Intensive Care Unit, Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China